CLINICAL TRIAL: NCT05510934
Title: Shared Care Thyroid Cancer Follow-up Utilizing Thyroid Cancer Assessment Reminder System (TCARS) Study - A Pilot Study.
Status: Recruiting | Type: Observational
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Other Study IDs: TCARS-2022
Record Dates: First submitted 2022-07-29; First posted 2022-08-22 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Low Risk Differentiated Thyroid Cancer
Keywords: low risk DTC; Shared-care model; decentralized clinical trial (DCT); DTC; Thyroid Cancer; Feasibility Study
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Shared-care Group: The Shared-care Group will comprise of patients who are receiving long term follow-up care for their condition by their PCP.
  Interventions: Behavioral: Shared-care model
- Control Group: The Control Group will be made of patients who are receiving long term follow-up care for their condition of low-risk DTC at the Halifax Interdisciplinary Thyroid Oncology Clinic (ITOC).

INTERVENTIONS:
Behavioral: Shared-care model — A Shared care follow-up strategy involving patients, PCPs and specialists that uses an automated reminder system (TCARS).
  Groups: Shared-care Group

SUMMARY:
This study aims to assess the feasibility of a shared-care model for low-risk differentiated thyroid cancer (DTC) patients, primary care practitioners (PCPs) and the tertiary care center utilizing a digital health-based thyroid cancer assessment reminder system (TCARS) in Medable with an expedited referral to specialists for rapid assessment in case of a concern of recurrence.

DETAILED DESCRIPTION:
Low risk differentiated thyroid cancer (DTC) is being increasingly diagnosed and although its overall survival is excellent, lifelong follow-up is needed due to the risk of ongoing health challenges and the cancer recurring. While it is not feasible to follow this growing number of patients in specialist centers due to limited resources, recent studies have suggested that simply discharging them to their PCP is not ideal because many PCPs do not feel confident in managing various aspects of DTC. More importantly, a large number of patients in Nova Scotia do not have regular access to PCPs and are thus followed by walk-in clinics or nurse practitioners.The optimal approach would therefore be, to establish a shared care follow-up model including participation from patients, primary care practitioners (PCPs) and specialists.

In this study, the feasibility of a shared care follow-up strategy involving patients, PCPs and specialists that uses an automated reminder system will be tested. This strategy will be compared to standard specialist only follow-up. The study population comprises 60 low risk adult DTC patients who will be randomly allocated to either Shared-care or Control group on a 1:1 basis (30 patients each).

The main objectives of this study is to:

1. Develop a digital health-based thyroid cancer assessment reminder system alerting patients and PCPs of patients' forthcoming appointment and guidelines.
2. Establish an expedited referral pathway to tertiary care for rapid assessment of patients discharged to PCPs in case of a risk of recurrence.
3. Identify the feasibility of the Shared-care model.
4. Compare the completion of the clinical assessments between Shared-care and Control Groups.
5. Compare patient and provider satisfaction and acceptability between Shared-care and Control Groups.
6. Compare PCP confidence in dealing with DTC before and after study completion.

ELIGIBILITY:
Inclusion Criteria:

Adult (>18 years old) consenting patients being followed at the Halifax Interdisciplinary Thyroid Oncology Clinic (ITOC) meeting the following criteria:

* AJCC stage 1 DTC with no radiological or biochemical evidence of thyroid cancer with undetectable high sensitivity serum thyroglobulin (hsTG <0.06 mcg/L*);
* Anti-thyroglobulin antibody (anti-TG AB <20 IU/ml*);
* Thyroid ultrasound scan [USS] negative for regional recurrence at least 24 months after most recent treatment;
* AJCC stage 2 DTC with no radiological or biochemical evidence of cancer (undetectable hsTG and anti-TG AB and negative thyroid USS) at least 48 months after most recent treatment
* Patient is comfortable with using the mobile or Medable application and has access to internet.

Exclusion Criteria:

Patient does not have a consented PCP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Control group = 30 patients, where 15 patients are from the Nova Scotia central zone, and 15 patients are from the Nova Scotia non-central zone.
  Shared-care group = 30 patients, where 15 patients are from the Nova Scotia central zone, and patients are from the Nova Scotia non-central zone .
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-09-30 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility outcomes | after up to 24 months (after the 2nd Follow-up)
  These outcomes will assess the feasibility of the pilot study. These include:
  * Number (%) of eligible patients who are approached for the study and agree to participate in either group.
  * Number (%) of eligible patients who are are approached for the study but refuse to participate in either group and reason for refusal.
  * Number (%) of patients who remain in the shared-care group at study end.
  * Number of patients who choose to terminate the study in either group and reason for termination.
  * Number of patients who lost their PCP and returned to specialist care.
DTC shared-care outcomes | after up to 24 months (after the 2nd Follow-up)
  These outcomes will be measured to compare shared-care vs control DTC patients during the study duration and prospectively entered into a computerized DTC outcome registry of all study patients to follow their progress. This will be separate from TCARS, which will contain no clinical information.This information will be entered by the study coordinator. These include:
  * Number (%) of patients having annual TG/anti-TG AB.
  * Number (%) of patients having annual neck ultrasound.
  * Number (%) of patients with TSH test every 6 months.
  * Number (%) of patients with TSH within target range and if outside target, whether thyroxine dose was adjusted and TSH rechecked.
  * Number (%) of patients with abnormal findings on neck ultrasound or TG/anti-TG AB test.
  * Number (%) of patients who were referred back to ITOC using the expedited referral sheet and reason for referral.

SECONDARY OUTCOMES:
Patient satisfaction outcomes | after up to 5 months (after 1st follow-up) and after up to 24 months (after 2nd follow-up)
  Patient satisfaction will be assessed in both groups using the Patient Satisfaction Questionnaire Short form (PSQ -18). The PSQ-18 is a Likert scale questionnaire, consisting of 18 items tapping each of the seven dimensions of satisfaction with medical care. These are 1) general satisfaction, 2) technical quality, 3) interpersonal manner, 4) communication, 5) financial aspects, 6) time spent with doctor, and 7) accessibility and convenience.
Patient and provider acceptability and experience outcomes | after up to 24 months (after 2nd Follow-up)
  Patient and provider satisfaction, acceptability and experience will be assessed through qualitative data gathered by provider (Specialist and PCP) interviews (n=8) and patient focus groups (n=12-16; 2 groups of 6-8 participants each).
PCP confidence in DTC management outcomes | after up to 5 months (after 1st follow-up) and after up to 24 months (after 2nd follow-up)
  PCP involvement and confidence in DTC management outcomes will be based on previously published surveys.
  The survey is based on the National Cancer Institute Survey of Physician Attitudes Regarding the Care of Cancer Survivors which was modified for thyroid cancer. In addition to the standard survey items, PCPs will be asked to report how confident they are in discussing key aspects of follow-up care with thyroid cancer survivors including:
  * Role of serum hsTG and anti-TG AB in long term surveillance.
  * Role of neck US in long term surveillance.
  * When to end long term surveillance.
  * When to refer back to specialist. All responses will be on a 5-point Likert type not at all confident to very confident.

OTHER OUTCOMES:
DCT (Medable) specific outcomes | after up to 5 months (after 1st follow-up) and after up to 24 months (after 2nd follow-up)
  Feedback on the use of the Medable (DCT) system will be assessed using qualitative data gathered through patient and PCP surveys. Some responses will be on a 5-point Likert-type scale from strongly disagree to strongly agree or very unlikely to likely. Other questions will be in a multiple choice format. An open dialogue box will appear at the end of the survey for respondents to enter additional comments.

CONTACTS AND LOCATIONS:
Overall Officials: Syed A. Imran, Dr., Principal Investigator — Nova Scotia Health
Locations (1):
- Nova Scotia Health, Halifax, Nova Scotia, Canada